CLINICAL TRIAL: NCT04589325
Title: The Effect of Anti-IL17 in New-onset Type 1 Diabetes: a Randomized, Double-blind, Placebo-controlled Trial
Brief Title: Ixekizumab Diabetes Intervention Trial (I-DIT)
Acronym: I-DIT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDIT001
Record Dates: First submitted 2020-09-24; First posted 2020-10-19 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Type1 Diabetes Mellitus
Keywords: Type 1 diabetes; New-onset; MMTT; Ixekizumab
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — ixekizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ixekizumab (Experimental)
  Interventions: Drug: Ixekizumab
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ixekizumab — Ixekizumab will be available at a concentration of 80 mg solution for injection in pre-filled syringes.
  Ixekizumab will be administrated by the patient via subcutaneous (s.c.) injections for a total treatment period of 12 months. Two s.c. injections (160 mg) will be administrated at week 0, one dose (80 mg) at week 2, 4, 6, 8, 10 and 12 and continue with a maintenance dose (80 mg) every 4th week for a total treatment period of 12 months.
  Other Names: Taltz
  Arms: Ixekizumab
Drug: Placebo — Placebo will be available at a concentration of 80 mg solution for injection in pre-filled syringes.
  Placebo will be administrated by the patient via subcutaneous (s.c.) injections for a total treatment period of 12 months. Two s.c. injections (160 mg) will be administrated at week 0, one dose (80 mg) at week 2, 4, 6, 8, 10 and 12 and continue with a maintenance dose (80 mg) every 4th week for a total treatment period of 12 months.
  Arms: Placebo

SUMMARY:
Although the clinical onset of type 1 diabetes (T1D) is acute, the progression of T1D occurs over many years often in a patchy manner with inflammation in certain lobes of the pancreas, leaving other lobes unaffected and long-lasting beta cells remain functional decades after diagnosis. Psoriasis share several aspects with T1D, e.g. the patchy inflammatory infiltrate consisting of tissue-resident memory (TRM) T cells, leaky blood vessels that facilitate leukocyte migration and the increased risk for systemic conditions. Moreover, interleukin (IL)-17 has shown to be increased in both persons with psoriasis and T1D. Activation of IL-17/IL-22 pathway is viewed to be both a hallmark of psoriasis and human T1D. Ixekizumab, an anti-IL17 biological agent, has shown marked therapeutic value in the treatment of subjects with psoriasis in several randomized trials and is currently an approved clinical therapy. Due to the many similarities in the current view of pathogenesis and manifestation of T1D and psoriasis it is possible that Ixekizumab can also influence the disease process of T1D.

DETAILED DESCRIPTION:
In this double-blind, placebo-controlled prospective trial, patients with newly diagnosed T1D will be randomized to receive either Ixekizumab or placebo in addition to their conventional therapy. The primary aim is to examine the effect of Ixekizumab on endogenous insulin production when administered to persons with newly diagnosed T1D. The planned study duration is 52 weeks with an extension phase for 3 years and includes 127 patients at 17 centers in Sweden. During the extension phase the participants will be examined during a visit after 1 and 3 years after the end of the study regarding insulin production (C-peptide and proinsulin secretion during a Mixed Meal Tolerance Test), glycaemic control, T1D auto-antibodies and insulin doses.

ELIGIBILITY:
INCLUSION CRITERIA:

* Signed informed consent and expected cooperation of the patients for the treatment and follow up must be obtained and documented according to ICH GCP, and national/local regulations before trial activities are begun.
* Must be willing and capable of taking the study drugs and meet for tests and follow up as described.
* Diagnosed Type 1 Diabetes (E10.9) within 100 days.
* First injection of insulin maximum 100 days prior to screening
* Aged 18-45 years old.
* Presence of antibodies at clinical practice or at screening to at least one of the following antigens: insulin/IAA, GAD-65, IA-2 and ZnT8.
* Remaining stimulated peak C-peptide ≥ 0.20 nmol/L. If age 36-45 years, peak C-peptide should be <2.0 nmol/L.
* Male subjects agree to use a reliable method of birth control during the study
* Female subjects:

Participants of childbearing age or childbearing potential who are sexually active who test negative for pregnancy must be counseled and agree to use either 1 highly effective method of contraception or 2 acceptable methods of contraception combined for the duration of the study and for at least 12 weeks following the last dose of study drug or remain abstinent during the study and for at least 12 weeks following the last dose of study drug.

If the highly effective contraceptive methods are contraindicated or strictly declined by patient, acceptable birth control methods may be considered. These may include combination of both of the following methods:

* Male or female condom with spermicide
* Cap, diaphragm, or sponge with spermicide

  1. Highly effective methods of contraception (use 1 form):

     1. combined oral contraceptive pill and mini-pill
     2. NuvaRing®
     3. implantable contraceptives
     4. injectable contraceptives (such as Depo-Provera®)
     5. intrauterine device (such as Mirena® and ParaGard®)
     6. contraceptive patch-ONLY women <198 pounds or 90 kg
     7. abstinence from sex
     8. vasectomy-for men in clinical studies
  2. Effective methods of contraception (use 2 forms combined)
* male condom with spermicide
* female condom with spermicide
* diaphragm with spermicide
* cervical sponge
* cervical cap with spermicide

Females who are not of childbearing potential include those who have undergone or who have:

* female sterilization
* hysterectomy
* menopause
* Müllerian agenesis (Mayer-Rokitansky-Küster-Hauser syndrome [also referred to as congenital absence of the uterus and vagina])

EXCLUSION CRITERIA:

* Contraindications to Ixekizumab.
* Treatment with any oral or injected glucose-lowering agents other than insulin.
* A history of haemolytic anaemia or significantly abnormal haematology/coagulation results at screening.
* Participation in other clinical trials with a new chemical entity within the previous 3 months.
* Subjects with severe obesity (BMI >35 kg/m2 if age 18-35 years and BMI >30 kg/m2 if age 36-45).
* Subjects with other autoimmune disease, e.g. Mb Crohn, Ulcerative colitis, Graves disease, psoriasis, psoriasis arthritis and axial spondylarthrosis, except celiac disease and hypothyroidism which do not need to be excluded for.
* Active serious or chronic infections (ie: in case patient had a serious infection (eg pneumonia, cellulitis), has been hospitalized, has received intravenous antibiotics for an infection within 12 weeks prior to screening visit, had a serious bone or joint infection within 24 weeks before screening visit, has ever had an infection of an artificial joint
* Known immunodeficiency or patient is immunocompromised to an extent that participation in the study would pose and unacceptable risk to the patient
* Tuberculosis
* History of HIV, hepatitis B or C
* Active or recurrent fungal infection
* Subjects with myocardial infarction, stroke, unstable angina or heart failure last 6 months
* Current clinically significant cardiac arrhythmias as verified by ECG
* Planned surgery during the treatment period of the study (except minor surgery on skin lesions, e.g., nevus)
* For female subjects: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 3- months after discontinuation.
* For male subjects: intent to procreate during the duration of the study or within 3 months after discontinuation or unwillingness of their partner to use effective contraceptive measures for the duration of the study and 4 months after discontinuation.
* Any history of malignancy the last 5 years except for completely resected squamous or basal cell carcinoma of the skin.
* Administration of live attenuated vaccine(s) (LAV) within 2 months of enrolment. Or intended use of LAV during the treatment period.
* The investigator judges that the clinical diagnosis of T1D set is incorrect or uncertain (needs to be confirmed by discussion with experienced diabetologist if excluding due to this criterion)
* Allergy against ingredients of the investigational products.
* Known allergy or hypersensitivity to any biologic therapy (active substance or excipients) that would pose an unacceptable risk to the patient if participating in the study
* Presence of serious disease or condition, which in the opinion of the investigator makes the patient non-eligible for the study.
* Liver injury criteria: patients with active hepatobiliary diseases or at screening having alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2.5 times the upper limit of normal (>2.5 x ULN)
* Laboratory abnormalities at screening:

  1. Neutrophil count < 1,500 cells/ μL (=1,5 *109 cells/ L)
  2. Platelet count < 100,000 cells/ μL (= 100 *109 cells/ L)
  3. Hemoglobin < 8.5 g/dL (= <85 g/L) (males) and <8g/dL (= <80 g/L) (women)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 127 (Estimated)
Dates: Start 2022-11-09 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Residual insulin secretion | 12 months
  Change in residual insulin secretion measured by stimulated C-peptide two-hour area under the curve profile measured by Mixed Meal Tolerance Test (MMTT) between baseline and week 52.

SECONDARY OUTCOMES:
Mean Insulin dosage per kilo bodyweight for 24 hours | 12 months
  Change in mean Insulin dosage per kilo bodyweight for 24 hours from baseline to week 52.
Time with glucose levels in range (3.9-10 mmol/L) | 12 months
  Change in time with glucose levels in range (3.9-10 mmol/l) measured by CGM/FGM from baseline to week 52.
Time in hypoglycaemia (<3.9 mmol/L) | 12 months
  Change in time in hypoglycaemia (<3.9 mmol/L) measured by CGM/FGM from baseline to week 52.
HbA1c | 12 months
  Difference in HbA1c from baseline to week 52.

OTHER OUTCOMES:
Time in hypoglycaemia (<3.0 mmol/L) | 12 months
  Change in time in hypoglycaemia (<3.0 mmol/L) measured by CGM/FGM from baseline to week 52.
Proinsulin/c-peptide ratio in serum as a measure of beta cell stress | 12 months
  Change in proinsulin/c-peptide ratio in serum as a measure of beta cell stress from baseline to week 52.
Time in target (3.9-8 mmol/L) | 12 months
  Change in time in target (3.9-8 mmol/L) measured by CGM/FGM from baseline to week 52.
Time in hyperglycaemia >10 mmol/L and ≥ 14 mmol/L | 12 months
  Change in time in hyperglycaemia >10 mmol/L and ≥ 14 mmol/L measured by CGM/FGM from baseline to week 52.
Glycaemic variability (mean amplitude of glycemic excursions (MAGE)) | 12 months
  Change in glycaemic variability measured by mean amplitude of glycemic excursions (MAGE) by CGM/FGM from baseline to week 52.
Glycaemic variability (coefficient of variation (CV)) | 12 months
  Change in glycaemic variability measured by coefficient of variation (CV) by CGM/FGM from baseline to week 52.
Glycaemic variability (standard deviation (SD)) | 12 months
  Change in glycaemic variability measured by standard deviation (SD) by CGM/FGM from baseline to week 52.
Proportion of patients with peak residual insulin secretion | 12 months
  Change in proportion of patients with peak residual insulin secretion measured by MMTT: stimulated C-peptide >0.4 pmol/mL from baseline to week 52
Change in World Health Organization-5 (WHO-5) scores from baseline and week 52. | 12 months
  Score 0 to 100; higher value indicates better well-being
Change in Diabetes Treatment Satisfaction Questionnaire (DTSQ) scores from baseline and week 52. | 12 months
  Score 0 to 36; higher value indicates better satisfaction and change in satisfaction (score -18 to 18; higher value indicates better change in satisfaction).
Change in Hypoglycaemia Fear Survey (Swe-HFS) scores from baseline and week 52. | 12 months
  Score 0 to 4; higher value indicates greater fear.
Change in Problem Areas in Diabetes Scale (PAID) scores from baseline and week 52. | 12 months
  Score 0 to 100; higher value indicates greater problems.
Change in International Physical Activity Questionnaire (IPAQ) scores from baseline and week 52. | 12 months
  Total Physical Activity Scores are calculated by Metabolic Energy Turnover (MET)-minutes/week score.

CONTACTS AND LOCATIONS:
Locations (17):
- Sweden (17):
  - Södra Älvsborg Hospital, Borås
  - Falu Lasarett, Falun
  - Sahlgrenska University Hospital, Sahlgrenska, Gothenburg
  - Sahlgrenska University Hospital, Östra Hospital, Gothenburg
  - Länssjukhuset Ryhov, Jönköping
  - Karlstad lasarett, Karlstad
  - Kristianstad Hospital, Kristianstad
  - Linköping University Hospital, Linköping
  - Lund University Hospital, Lund
  - Vrinnevi Hospital, Norrköping
  - Örebro University Hospital, Örebro
  - Skaraborgs sjukhus, Skövde
  - Centrum för Diabetes,, Stockholm
  - Södersjukhuset Hospital, Stockholm
  - NU-Hospital Group, Uddevalla
  - Uppsala Academic Hospital, Uppsala
  - Varbergs sjukhus, Varberg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Seyed Ahmadi S, Korsgren O, Jansson PA, Lind M. Design and methods of the Ixekizumab Diabetes Intervention Trial (I-DIT): protocol for a phase 2, randomised, multicentre, placebo-controlled, double-blind trial of anti-interleukin 17 as a treatment option for adults with new-onset type 1 diabetes. BMJ Open. 2025 Nov 12;15(11):e103486. doi: 10.1136/bmjopen-2025-103486. PMID 41224288